CLINICAL TRIAL: NCT06997458
Title: Clinical Implementation of Liquid Biopsy in Cancer Through Next Generation Sequencing (NGS) Panels in the Andalusian Public Health System
Brief Title: Liquid BiOpsy, Lung and Colon Cancer in AndaluciA
Acronym: LOLA-PROJECT
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Tempus AI (Industry)
Responsible Party: Principal Investigator, María José Serrano Fernández, Principal Investigator, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Other Study IDs: LCI2024-2027
Record Dates: First submitted 2025-04-25; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC)
Keywords: Liquid Biopsy; cfDNA; ctDNA; Metastatic Cancer; NGS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Streck tubes with 8.5mL of blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with radiologic evidence of metastatic (stage IV) NSCLC: * Patients diagnosed with the 8th Edition of the Tumor, Node, Metastasis (TNM) staging system for Lung Cancer approved by International Association for the Study of Lung Cancer (IASLC) and the American Joint Committee on Cancer (AJCC): IV (Any T, Any N, M1a-c)
  * Histologically confirmed NSCLC (adenocarcinoma)
  * Performance status of 0-2 (ECOG PS)
  * Estimated life expectancy ≥3 months
  * Treatment naïve patients (chemotherapy, immunotherapy, targeted therapy, radiotherapy).
  * Smokers or Non-Smokers
  Interventions: Diagnostic Test: xF Tempus assay
- Patients with radiologic evidence of metastatic (stage IV) CRC: * Patients diagnosed with the Tumor, Node, Metastasis (TNM) staging system for Colorectal Cancer approved by the American Joint Committee on Cancer (AJCC): IV (Any T, Any N, M1a-c).
  * Histologically confirmed CRC (adenocarcinoma).
  * Performance status of 0-2 (ECOG PS)
  * Estimated life expectancy ≥3 months
  * Treatment naïve patients (chemotherapy, immunotherapy, targeted therapy, radiotherapy).
  Interventions: Diagnostic Test: xF Tempus assay

INTERVENTIONS:
Diagnostic Test: xF Tempus assay — The blood will be collected and sent to Tempus Labs using the standard sample collection kit containing all the necessary elements to guarantee shipment to Tempus Labs. Two Streck tubes with 8.5mL of blood per tube will be sent to Tempus Labs.
  The ctDNA isolation and automatic library preparation will be performed using TEMPUS technology (Finkel et al 2021).
  The NGS analyses will be developed using the xF Tempus assay. This assay involves a panel with hybrid gene capture that detects actionable oncologic targets in four variant classes: single-nucleotide variants (SNVs), insertions/deletions (indels), copy number variants (CNVs), and gene rearrangements. The NGS sequencing is performed using NovaSeq 6000Dx Sequencing System (Illumina, Inc) equipment, according to Tempus protocols. (Finkel et al 2021).

SUMMARY:
The objective of the LOLA Project is to analyse the impact of adopting xF liquid biopsy panel, in the real world of the Andalusian Health Public System in terms of impact on clinical practice and cost through the assessment of clinical impact, duration of turnaround time (TAT) of xF test vs standard of care and the analysis of resource utilisation.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* More than 18 years old
* Both genders
* Ability to provide written informed consent

Specific criteria:

* NSCLC

  * Patients diagnosed with the 8th Edition of the Tumor, Node, Metastasis (TNM) staging system for Lung Cancer approved by International Association for the Study of Lung Cancer (IASLC) and the American Joint Committee on Cancer (AJCC): IV (Any T, Any N, M1a-c)
  * Histologically confirmed NSCLC (adenocarcinoma)
  * Performance status of 0-2 (ECOG PS) ○ Estimated life expectancy ≥3 months
  * Treatment naïve patients (chemotherapy, immunotherapy, targeted therapy, radiotherapy).
  * Smokers or Non-Smokers
* CRC

  * Patients diagnosed with the Tumor, Node, Metastasis (TNM) staging system for Colorectal Cancer approved by the American Joint Committee on Cancer (AJCC): IV (Any T, Any N, M1a-c)
  * Histologically confirmed CRC (adenocarcinoma)
  * Performance status of 0-2 (ECOG PS)
  * Estimated life expectancy ≥3 months
  * Treatment naïve patients (chemotherapy, immunotherapy, targeted therapy, radiotherapy).

Exclusion Criteria:

* General: History of any other cancer within the previous 5 years, except non-melanoma skin cancer
* General: Absence of Informed consent. > Pregnant or nursing women. > Small cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic adenocarcinoma (NSCLC: 250 and CRC: 250)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
To analyse the impact of adopting large (TEMPUS) NGS panels in the real world of the Andalusian Health Public System in terms of impact on clinical practice and cost. | through study completion, an average of 3 year
  Proportion of patients with at least one actionable variant (%)

CONTACTS AND LOCATIONS:
Overall Officials: M Jose Serrano, PhD, Principal Investigator — Centre for Genomics and Oncological Research - Pfizer - University of Granada - Andalusian Regional Government (GENyO) & University Hospital Virgen de la Nieves; Valeria Denninghoff, PhD, Study Director — Centre for Genomics and Oncological Research - Pfizer - University of Granada - Andalusian Regional Government (GENyO)
Locations (1):
- Centre for Genomics and Oncological Research - Pfizer - University of Granada - Andalusian Regional Government (GENyO), Granada, Andalusia, Spain

REFERENCES:
- [Background] Rolfo C, Cardona AF, Cristofanilli M, Paz-Ares L, Diaz Mochon JJ, Duran I, Raez LE, Russo A, Lorente JA, Malapelle U, Gil-Bazo I, Jantus-Lewintre E, Pauwels P, Mok T, Serrano MJ; ISLB. Challenges and opportunities of cfDNA analysis implementation in clinical practice: Perspective of the International Society of Liquid Biopsy (ISLB). Crit Rev Oncol Hematol. 2020 Jul;151:102978. doi: 10.1016/j.critrevonc.2020.102978. Epub 2020 May 5. PMID 32428812
- [Background] Rolfo C, Denninghoff V. Globalization of precision medicine programs in lung cancer: a health system challenge. Lancet Reg Health Eur. 2023 Dec 12;36:100819. doi: 10.1016/j.lanepe.2023.100819. eCollection 2024 Jan. No abstract available. PMID 38170059
- [Background] Pisapia P, Costa JL, Pepe F, Russo G, Gragnano G, Russo A, Iaccarino A, de Miguel-Perez D, Serrano MJ, Denninghoff V, Quagliata L, Rolfo C, Malapelle U. Next generation sequencing for liquid biopsy based testing in non-small cell lung cancer in 2021. Crit Rev Oncol Hematol. 2021 May;161:103311. doi: 10.1016/j.critrevonc.2021.103311. Epub 2021 Mar 26. PMID 33781866
- [Background] Finkle JD, Boulos H, Driessen TM, Lo C, Blidner RA, Hafez A, Khan AA, Lozac'hmeur A, McKinnon KE, Perera J, Zhu W, Dowlati A, White KP, Tell R, Beaubier N. Validation of a liquid biopsy assay with molecular and clinical profiling of circulating tumor DNA. NPJ Precis Oncol. 2021 Jul 2;5(1):63. doi: 10.1038/s41698-021-00202-2. PMID 34215841
- [Background] Malapelle U, Pisapia P, Addeo A, Arrieta O, Bellosillo B, Cardona AF, Cristofanilli M, De Miguel-Perez D, Denninghoff V, Duran I, Jantus-Lewintre E, Nuzzo PV, O'Byrne K, Pauwels P, Pickering EM, Raez LE, Russo A, Serrano MJ, Gandara DR, Troncone G, Rolfo C. Liquid biopsy from research to clinical practice: focus on non-small cell lung cancer. Expert Rev Mol Diagn. 2021 Nov;21(11):1165-1178. doi: 10.1080/14737159.2021.1985468. Epub 2021 Oct 11. PMID 34570988
- See also: Centre for Genomics and Oncological Research - Pfizer - University of Granada - Andalusian Regional Government (GENyO) — https://www.genyo.es/
- See also: Public Procurement of Innovation: Liquiq Biopsy — https://www.liquidbiopsyproject.com/es
- See also: Andalusian Health System — https://www.sspa.juntadeandalucia.es/servicioandaluzdesalud/